CLINICAL TRIAL: NCT04908306
Title: IMAGE-HF: Project IIa - Canadian CArdiomyopathy Registry for Device Therapy (CanCARD-MR)
Brief Title: IMAGE-HF: Project IIa Canadian CArdiomyopathy Registry for Device Therapy
Acronym: CanCARD-MR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: 2011308-01
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Delayed enhanced MRI in patients (of either ischemic or non-ischemic cause) being referred for primary prevention ICD

DETAILED DESCRIPTION:
Device therapy using defibrillators and cardiac resynchronization therapy (CRT) is an important advance in the care of patients with acquired heart disease and heart failure. In specific groups these devices appear to significantly reduce the risk of sudden cardiac death and progression of heart failure. However, our ability to identify ideal candidates, and those who are most likely to respond and benefit from this therapy, is poor.

Preliminary studies using specialized Magnetic Resonance Imaging (MRI) appears to be one of the more valuable ways of predicting response to device therapy and holds substantial promise for patients with cardiomyopathy.

Large, prospective registries are necessary to explore its real-world utility for risk prediction across a broad spectrum of patients. Can-CARD MR is a national, multi-centre registry designed to address this particular need.

ELIGIBILITY:
Inclusion Criteria:

* .Any patient accepted for primary prevention ICD (+/-) CRT)

Exclusion Criteria:

* Known contra-indications to MRI.
* Recent myocardial infarction or revascularization procedure within the past 3 months.
* GFR (glomerular filtration rate) ≤ 30 ml. / min/ m2.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred for or being considered for primary prevention ICD, with or without CRT, will be recruited from the Electrophysiology services at each enrolling site
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2011-10-11 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a)appropriate ICD therapy (shock or anti-tachycardia pacing (ATP)) or sudden cardiac death | 1 year
  Occurrence of a)appropriate ICD therapy (shock or anti-tachycardia pacing (ATP)) or sudden cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: David Birnie, Principal Investigator — Ottawa Heart Institute Research Corporation